CLINICAL TRIAL: NCT06609096
Title: The Effect of Sexual Counselling Based on PLISSIT and BETTER Model on Sexual Function and Quality of Sexual Life After Hysterectomy: A Randomised Controlled Trial
Brief Title: The Effect of Sexual Counselling Based on PLISSIT and BETTER Model After Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Sevil Cicek Ozdemir, Assistant professor, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 908520
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Hysterectomy; PLISSIT Model; Sexual Health Quality of Life; Sexual Function; Sexual Health
Keywords: sexual health; Hysterectomy; Sexual Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In order to prevent outcome reporting bias, the data obtained from the study will be coded as A, B and C by an independent researcher and transferred to the SPSS program. Group assignment will be concealed from the researchers during the data analysis and reporting process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PLISSIT Group (Experimental): Women assigned to the sexual counseling group based on the PLISSIT model will receive four sessions in total, once a week. Each session consisted of an average of 30 min. Sessions will be conducted online as individual counselling sessions. The Plissit model was used based on a four-stage approach. These stages are (P-Permission): Permission, (Ll- Limited Information), providing limited information (SS-Specific Suggestions): Giving specific suggestions, (IT- Intensive Therapy): Intensive Therapy. In this study, the first three stages of the model will be applied. After the first three stages of the model are implemented, women with ongoing sexual problems are referred to specialized sexual therapists for intensive treatment/therapy.
  Interventions: Behavioral: Sexual counseling based on the PLISSIT model
- BETTER Group (Experimental): Women assigned to the sexual counseling group based on the BETTER model will receive four sessions in total, once a week. Each session will consist of 30 minutes on average. Better model consists of Bring up the topic, Explain, Telling, Timing, Education and Recording steps. The sessions will be conducted online as individual counselling sessions.
  Interventions: Behavioral: Sexual counseling based on the BETTER model
- Control Group (No Intervention): Women in the control group will not receive any intervention.

INTERVENTIONS:
Behavioral: Sexual counseling based on the PLISSIT model — Four sessions of sexual counseling based on the PLISSIT model will be provided. The intervention consisted of four consecutive sessions, with one session per week. Each session is 30 minutes on average.
  Arms: PLISSIT Group
Behavioral: Sexual counseling based on the BETTER model — A total of four sessions of sexual counseling based on the BETTER model will be provided. The intervention consists of four consecutive sessions, one session per week. Each session is 30 minutes on average.
  Arms: BETTER Group

SUMMARY:
Sexuality is affected by several physiological, cultural, social, and psychological factors. Hysterectomy is one of the factors that affects sexuality. Evidence suggests that hysterectomy, affects the sexual function of women. Therefore, this study aimed to evaluate the effect of sexual counseling based on the PLISSIT and BETTER models on sexual function and quality of sexual life of women after hysterectomy. This study is a randomized controlled trial with a three-arm parallel design. One of the experimental groups will receive sexual counseling based on the PLISSIT model and the other will receive sexual counseling based on the BETTER model. The control group will not receive any intervention. The difference between the intervention groups and the control group will be evaluated.

DETAILED DESCRIPTION:
Nurses are integral members of the health care team in providing care and counseling for sexual health. The provision of education and counseling services to enhance sexual health and research on the subject play significant roles for nurses. In this context, nurses should facilitate up-to-date information dissemination to clients by investigating sexual counseling models. Furthermore, nurses have crucial duties and responsibilities for maintaining evidence-based care practices that utilize these models. Addressing sexual life and adopting a holistic approach to nursing care services are essential considerations. The utilization of models is recommended to assist nurses in evaluating sexuality of patients, which is a sensitive subject, in an appropriate manner and to provide them with the most suitable care in this regard. One such model was the PLISSIT Model. The PLISSIT Model was employed to assess and improve sexual health in patients with breast cancer, multiple sclerosis, gynecologic cancer, type 2 diabetes mellitus, HIV-positive status, and stoma. Additionally, it is actively used in different life stages of women such as pregnancy and postpartum period. In the literature, the results of studies in which sexual counseling based on the PLISSIT model was applied to women undergoing hysterectomy indicate that the model has positive effects on sexual function and quality of sexual life. However, the PLISSIT model has limitations, such as the requirement for skills at the fourth stage of sexual rehabilitation at the 4th stage and its linearity (progressing from one level to another). One of the alternative approaches in sexual counseling is the BETTER Model due to its specific emphasis on developing dialogues on sexual health and the importance of sexual issues. This model has been utilized in the literature to provide sexual counseling to women with multiple sclerosis, women with breast cancer, infertile women, and postpartum women. However, no study was identified in the literature in which sexual counseling based on the BETTER model was provided to women with hysterectomy. Evidence of the effectiveness of model-based sexual counseling in women with sexual dysfunction after hysterectomy is insufficient.

ELIGIBILITY:
Inclusion Criteria:

* Having a sexual partner
* Sexual intercourse within the last month,
* A score below 26.55 on the Female Sexual Function Scale,
* At least 3 months after the hysterectomy operation,
* No previous radiotherapy or chemotherapy treatment,
* Not having any communication problems (mental, auditory, visual, etc.),
* Not being involved in any other sexuality-related treatment program,
* Becoming literate,
* Having a smartphone,
* Access to the Internet
* Volunteering to participate in the study

Exclusion Criteria:

* Different treatment protocols due to malignancy (radiotherapy and chemotherapy or additional surgical treatment of the reproductive organs)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female participants who have had a hysterectomy operation can participate in this study.
Enrollment: 52 (Actual)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Sexual Quality of Life Scale-Female Scale | Change from baseline level sexual function to month 1 and month 2
  Sexual Quality of Life Scale-Female (SQOL-F) developed by Symonds et al. (2005). The scale should be completed by considering sexual life in the last four weeks. The scale consisted of 18 items and was evaluated between 1 and 6 points. As the scale score increased, so did the quality of sexual life.
Female Sexual Function Scale | Change from baseline level sexual function to month 1 and month 2
  The Female Sexual Function Scale (FSFI) developed by Rosen et al. (2000) focused on sexual problems in the last four weeks and evaluated sexual function. It consists of 19 questions and six sub-dimensions including desire, arousal, lubrication, orgasm, satisfaction, and pain. The scores obtained from the scale varied between 2 and 36. As the scale score increased, sexual function also increased. The cutoff score of the scale was 26.55. Those with a score of 26.55 and below were considered to have female sexual dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Sevil Çiçek Özdemir, Asst. Prof., Principal Investigator — Kütahya Health Sciences University
Locations (2):
- Turkey (Türkiye) (2):
  - Gazi University Health Research And Application Center, Ankara
  - Kütahya Health Sciences University, Kütahya

IPD SHARING:
Plan to Share IPD: No
There are no plans to make individual participant data available to other researchers.